CLINICAL TRIAL: NCT07212686
Title: An Open-Label, Single-Center Study of Synthetic Angiotensin II/Giapreza in Pediatric Patients With Refractory Hypotension Despite Receiving Fluid Therapy and Vasoactive Therapy
Brief Title: Synthetic Angiotensin II/Giapreza in Pediatric Patients With Refractory Hypotension
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Todd Sweberg (Other)
Collaborators: Innoviva Specialty Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Todd Sweberg, MD, Northwell Health
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0641-CCMC
Record Dates: First submitted 2025-06-16; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Vasodilatory Shock
Keywords: Vasodilatory shock; Angiotensin II; Pediatric Critical Care Medicine
MeSH Terms: interventions — Angiotensin I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pediatric patients in vasodilatory shock (Experimental): Patients enrolled in the study who meet inclusion criteria will receive Angiotensin-II per the titration protocol.
  Interventions: Drug: Angiotensin-II

INTERVENTIONS:
Drug: Angiotensin-II — Angiotensin-II will be given per the titration protocol.

SUMMARY:
The goal of this clinical trial is to determine the safety and efficacy of Angiotensin-II in the treatment of pediatric patients in fluid refractory vasodilatory shock. The main questions it aims to answer are:

* To evaluate the change in blood pressure or reduction of vasoactive requirements (norepinephrine equivalent dosing) after initiating Angiotensin II
* To establish the safety and tolerability of Angiotensin-II in pediatric patients Participants will receive Angiotensin-II in addition to standard of care therapy for vasodilatory shock.

  * The study team will then monitor the patient's vital signs, blood work, and for any potential side effects from the drug.
  * An ultrasound will be performed to look at blood flow through the kidney in the setting of vasodilatory shock.
  * A follow up phone call to check in with the patient will be performed 28 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients less than 18 years of age who have received at least 40 mL/kg of crystalloid or colloid equivalent fluid resuscitation for vasodilatory shock
* Titration of standard of care vasoactive medications for a minimum of 2 hours with persistent refractory hypotension for age, and who require a total sum NE equivalent dose of > 0.1 μg/kg/min for a minimum of 1 hours and a maximum of 24 hours prior to initiation of Angiotensin-II.
* Indwelling arterial and central venous lines.
* Parent or legal guardian is willing and able to provide informed consent and assist the patient in complying with all protocol requirements.

Exclusion Criteria:

* Standing DNR/DNI order
* Alternative shock diagnosis i.e. cardiogenic shock or post cardiac surgery
* Cannulated to extracorporeal membrane oxygenation
* Pre-existing condition confounding outcome determination such as terminal illness
* Patients diagnosed with acute occlusive coronary syndrome requiring pending intervention.
* Patients who have a history of asthma or are currently experiencing bronchospasm requiring the use of inhaled bronchodilators and who are not mechanically ventilated.
* Patients with acute mesenteric ischemia or a history of mesenteric ischemia.
* Patients with active bleeding AND an anticipated need of multiple transfusions (within 48 hours of Screening).
* Patients with active bleeding, hemoglobin < 7 g/dL, or any other condition that would contraindicate serial blood sampling.
* Patients requiring more than 5 mg/kg daily of hydrocortisone or equivalent glucocorticoid medication as a standing dose.
* Patients with an expected lifespan of < 12 hours or withdrawal of life support within 24 hours of screening.
* Patients currently using an angiotensin converting enzyme inhibitor or angiotensin receptor blocker.
* Patients with a known allergy to mannitol.
* Patients who are currently participating in another investigational clinical trial.
* Patients of childbearing potential who are known to be pregnant at the time of screening.
* Prisoners
* Patient's with Raynaud phenomenon, systemic sclerosis, or vasospastic disease.

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who have improvement in mean arterial pressure or reduction in sum norepinephrine equivalent at Hour 2 after the start of Synthetic Angiotensin-II | From enrollment to Hour 2
  Percentage (%) of patients who have improvement in mean arterial pressure (MAP, mmHg) or reduction in sum norepinephrine (NE) equivalent at Hour 2 after the start of Synthetic Angiotensin-II

SECONDARY OUTCOMES:
Change in MAP | From enrollment to 24 hours
  Change in mean arterial pressure (mmHg) from baseline to 24 hours
Change in systolic blood pressure | From enrollment to 24 hours
  Change in systolic blood pressure (mmHg) from baseline to 24 hours
Change in diastolic blood pressure | From enrollment to 24 hours
  Change in diastolic blood pressure (mmHg) from baseline to 24 hours
Change in concentration of serum lactate | From enrollment to 24 hours
  Change in concentration of serum lactate (mmol/L) from baseline to 2 hours
Change in pSOFA score | From enrollment to 24 hours
  Change in pSOFA score from screening to 24 hours (%)
Change in PRSIM-III score | From enrollment to 24 hours
  Change in PRSIM-III score from screening to 24 hours (%)
Change in total neutrophil count | From enrollment to 24 hours
  Change in total neutrophil count (cells/µL) from the start of Synthetic Angiotensin-II to 24 hours
Change in renal resistive index (%) | From enrollment to 24 hours
  Change in renal resistive index (%) from the start of Synthetic Angiotensin-II to 24 hours after the start of Synthetic Angiotensin-II

OTHER OUTCOMES:
Change in tissue oxygenation over 2 hours | From enrollment to Hour 2
  Change in tissue oxygenation as defined by peripheral oxygen saturation (%) from baseline to 2 hours
Change in tissue oxygenation over 24 hours | From enrollment to Hour 24
  Change in tissue oxygenation as defined by peripheral oxygen saturation (%) from baseline to 24 hours
Change in heart rate | From enrollment to Hour 2
  Change in heart rate (beats per minute) from baseline to 2 hours
Change in sum norepinephrine equivalent dose over 24 hours | From enrollment to 24 hours
  Change in sum norepinephrine equivalent dose (μg/kg/min) from baseline to 24 hours
28-day all-cause mortality | From enrollment to Day 28
  28-day all-cause mortality (%)
Number of ventilator days | From enrollment to Day 28
  Number of ventilator days
Ventilator free days | From enrollment to Day 28
  Number of ventilator free days
Days on vasoactive support | From enrollment to Day 28
  Number of days on vasoactive support
Change in T cell cell count | From enrollment to Day 28
  Change in T cell cell count (cells/µL)
Change in in serum cytokine levels | From enrollment to Day 28
  Change in in serum cytokine levels over time (pg/dL)
Change in renal resistive index (%) over time | From enrollment to 28 days
  Change in renal resistive index (%) over time
Change in renal blood flow over time | From enrollment to 28 days
  Change in renal blood flow (mL/min) over time
Change in power doppler by point of care ultrasound assessment | From enrollment to 28 days
  Change in power doppler by point of care ultrasound assessment (AU)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cohen Children's Medical Center of Northwell Health, New Hyde Park, New York
  - Cohen Children's Medical Center, Queens, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey DM, Chima RS, Tidmarsh GF, Williams MD. Synthetic Human Angiotensin II in Pediatric Patients With Vasodilatory Shock: A Report on Two Patients. Crit Care Explor. 2019 Aug 15;1(8):e0036. doi: 10.1097/CCE.0000000000000036. eCollection 2019 Aug. PMID 32166277
- [Background] Tezel O, Hutson TK, Gist KM, Chima RS, Goldstein SL, Stanski NL. Utilization of Synthetic Human Angiotensin II for Catecholamine-Resistant Vasodilatory Shock in Critically Ill Children: A Single-Center Retrospective Case Series. Crit Care Explor. 2023 Sep 12;5(9):e0978. doi: 10.1097/CCE.0000000000000978. eCollection 2023 Sep. PMID 37711646
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561